CLINICAL TRIAL: NCT02387320
Title: Evaluation of a Self-Care Toolkit in Surgical Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: San Antonio Military Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 396717
Record Dates: First submitted 2014-11-17; First posted 2015-03-13 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Anxiety; Pain; Nausea; Fatigue; Sleep Disturbance
Keywords: Anxiety; Pain; Nausea; Fatigue; Sleep Disturbance; Breast Cancer; Surgery
MeSH Terms: conditions — Anxiety Disorders; Pain; Nausea; Fatigue; Parasomnias; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Care Toolkit (Experimental): Women randomized to self-care toolkit group will receive a toolkit which includes a spiral-bound instruction manual, a section of the manual that can be used as a journal, a portable mp3 player with 8 audiofile tracks with guided meditations to reduce stress and anxiety, and two acupressure wristbands to help prevent nausea.
  Interventions: Other: Self-Care Toolkit
- Standard Care (No Intervention): Women randomized to the standard care group will be informed that they will continue to receive standard of care as delivered by the SAMMC Oncology Department. The research team will inform women randomized to standard care that they will receive the self-care toolkit at their two week post-operative visit and will be able to use it subsequently if they choose to.

INTERVENTIONS:
Other: Self-Care Toolkit — The self-care toolkit was designed and created for individuals undergoing surgery and/or invasive medical procedures. It provides individuals with guided instruction to learn several evidence-informed mind-body skills (e.g., breathing, relaxation, meditation, guided imagery) and tools (e.g., acupressure wristbands, journal) in order to regulate their own physiologic and emotional reactions to stressful situations and to lessen symptoms associated with surgery (principally pain, anxiety, nausea, fatigue, sleep disturbance).
  Arms: Self-Care Toolkit

SUMMARY:
This randomized controlled trial (RCT) in newly-diagnosed breast cancer patients seeks to determine the effectiveness of a self-care toolkit on specific symptoms associated with surgery as compared to a standard care group.

DETAILED DESCRIPTION:
The main research questions focus on whether the toolkit provides short-term benefits on symptoms associated with surgery (i.e., pain, anxiety, nausea) and whether it impacts emotional distress and other symptoms (i.e., pain, fatigue, sleep disturbance, global health, quality of life) at a two-week post-operative time point. This study will be conducted at San Antonio Military Medical Center (SAMMC) in active duty, veteran, and military dependent women newly diagnosed with breast cancer for whom surgery (e.g., lumpectomy or mastectomy) is the initial treatment option. One to two weeks prior to surgery, women diagnosed with breast cancer at SAMMC Oncology Department will be invited to participate in this study. Those who meet criteria and agree to participate will be enrolled on-study and randomly assigned to either the surgical toolkit group or standard care group. During the pre-operative period, women in the intervention group will be asked to read through the manual, listen to each of the 8 audiofiles at least once but as many times as desired, and to wear the acupressure wristbands during surgery. Women randomized to the standard care group will not receive an intervention prior to surgery but will receive the toolkit at study completion. The rationale for providing women in the standard care group with the toolkit at their post-operative visit is that the skills of breathing, meditation, and guided imagery might be potentially beneficial for them to use during their subsequent treatment or a future surgery. Additionally, qualitative interviews will be conducted in a cohort of women from the intervention group, at a two-week post-operative time point to assess their impressions and satisfaction with the toolkit; questions will focus on whether the individual used each of the toolkit's components, frequency of use, how she would rate the product's attributes (e.g., ease of use, clarity of instructions, quality rating, helpfulness), and perceptions about the helpfulness and usefulness of learned mind-body skills.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Women treated at SAMMC Oncology clinic or CRDAMC Oncology clinic for newly-diagnosed breast cancer for whom surgery (e.g., lumpectomy or mastectomy) is the initial treatment option

Exclusion Criteria:

* Women receiving chemotherapy, radiation or hormone therapy as first line treatment for breast cancer (i.e., any of these treatment options prior to surgery)
* Severe hearing-impairment (i.e., that would interfere with ability to hear the toolkit audiofiles)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change from preoperative in VAS General Anxiety at post-operative | Pre-operative (30 minutes to 5 hours prior to surgery) , Post-operative (within 10 hours after surgery)
  Anxiety is rated by the patient on a scale of 0 to 10, 0 being "not at all anxious" and 10 being "extremely anxious." This instrument will take up to 1 minute to complete.

SECONDARY OUTCOMES:
Change from pre-operative DVPRS at post-operative | Pre-operative (30 minutes to 5 hours prior to surgery) , Post-operative (within 10 hours after surgery)
  The Defense and Veterans Pain Rating Scale (DVPRS) is a graphic tool to facilitate self-reported pain rating from patients. The instrument uses a scale from 0-10, 0 being "no pain" to 10 being "as bad as it could be, nothing else matters." This instrument will take up to 1 minute to complete.
Change from preoperative VAS Nausea at post- operative | Pre-operative (30 minutes to 5 hours prior to surgery) , Post-operative (within 10 hours after surgery)
  Nausea is rated by the patient on a scale of 0 to 10, 0 being "no nausea" and 10 being "extreme nausea." This instrument will take up to 1 minute to complete.
Change from baseline (PROMIS-57) Fatigue to pre-operative and follow-up 2 weeks post-operative | Baseline, Pre-operative (30 minutes to 5 hours prior to surgery), follow-up 2 weeks post-operative
  The National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) profile measure (PROMIS-57) includes eight primary domains: anxiety, pain intensity, pain interference, fatigue, sleep disturbance, depression, physical function, and satisfaction with social roles. This instrument takes approximately 25 minutes to complete.
Change from baseline (PROMIS-57) Sleep Disturbance to pre-operative and follow-up 2 weeks post-operative | Baseline, Pre-operative (30 minutes to 5 hours prior to surgery), Follow-up 2 weeks post-operative
  The National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) profile measure (PROMIS-57) includes eight primary domains: anxiety, pain intensity, pain interference, fatigue, sleep disturbance, depression, physical function, and satisfaction with social roles. This instrument takes approximately 25 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly McConnell, EdD, Principal Investigator — Samueli Institute
Locations (2):
- United States (2):
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - San Antonio Military Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No